CLINICAL TRIAL: NCT00003605
Title: Rituximab Anti-CD20 Monoclonal Antibody Plus Oral Cyclophosphamide as Initial Treatment of Indolent Lymphoma
Brief Title: Rituximab Plus Cyclophosphamide in Treating Patients With Indolent Stage III or Stage IV Non-Hodgkin's Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no patient accrual
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Collaborators: Cancer Biotherapy Research Group (Other)
Responsible Party: Robert O. Dillman, MD, Hoag Memorial Hospital Presbyterian
Purpose: Treatment
Other Study IDs: CDR0000066680; CBRG-9801; GENENTECH-CBRG-9801; NBSG-9801; NCI-V98-1483
Record Dates: First submitted 1999-11-01; First posted 2004-08-04 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Lymphoma
Keywords: Waldenstrom macroglobulinemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy and monoclonal antibody therapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of rituximab plus cyclophosphamide in treating patients who have indolent stage III or stage IV non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity associated with cyclophosphamide and rituximab (IDEC-C2B8 monoclonal antibody) as first line treatment in patients with stage III or IV indolent B-cell lymphoma. II. Determine the objective tumor response rate and duration of response associated with this first line treatment in these patients. III. Determine the failure-free and overall survival for these patients. IV. Compare the response rate and survival rates for patients with indolent lymphoma who were treated with this treatment as the first systemic therapy for their disease with response rates and survival observed for similar patients treated in published trials. V. Determine the quality of life associated with this treatment in this patient population.

OUTLINE: This is an open label study. Patients receive oral cyclophosphamide daily and rituximab (IDEC-C2B8 monoclonal antibody) IV on days 1, 8, 15, and 22 for the first 4-week course. Patients then receive oral cyclophosphamide daily and rituximab IV monthly until 2 months beyond maximum response. Patients are treated for at least 6 months but no more than 18 months in the absence of disease progression. Patients are followed every 3 months for 2 years, then every 6 months for the next 2 years, and then annually for up to 10 years.

PROJECTED ACCRUAL: There will be 20-40 patients accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage III or IV indolent B-cell lymphoma Diffuse small cleaved cell lymphoma Follicular small cleaved cell lymphoma Follicular mixed cell lymphoma Follicular large cell lymphoma At least 1 lymph node or visceral lesion at least 2 cm in diameter

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Lymphocyte count less than 5,000/mm3 Hepatic: Not specified Renal: Not specified Other: No active infection No concurrent life threatening disease Not pregnant Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: No prior therapy for lymphoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1998-05; Primary Completion 2000-01 (Actual); Study Completion 2000-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert O. Dillman, MD, FACP, Study Chair — Cancer Biotherapy Research Group
Locations (3):
- United States (3):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Bloomington Hospital, Bloomington, Indiana
  - St. Joseph Regional Cancer Center, Bryan, Texas